CLINICAL TRIAL: NCT05546645
Title: Validation of a Questionnaire to Assess Bronchial Mucus Hypersecretion in Asthmatic Patients. Questionnaire "T-sec" (Secretion Test).
Brief Title: Development of "T-sec" Questionnaire
Acronym: T-sec
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-TSC-2022-09
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-03

CONDITIONS: Asthma
Keywords: Asthma; Hypersecretion; Sputum
MeSH Terms: conditions — Asthma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Hypersecretion questionnaire

SUMMARY:
To design and validate a questionnaire that allows objective assessment of the level of bronchial mucus hypersecretion.

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory disease associated with bronchial mucus hypersecretion (MBH) due to various mechanisms, such as increased mucin secretion, plasma exudation and cytokines. It is currently known that MBH in asthmatic patients is associated with increased mortality and reduced pulmonary function, but there is no tool for its objective assessment.

The aim of the study is to design and validate a questionnaire to objectively assess the level of bronchial mucus hypersecretion in patients with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 30 and 99 years
* Clinical diagnosis of asthma

Exclusion Criteria:

* Non-Spanish-speaking patients
* Inability to complete the questionnaires
* Failure to sign the informed consent form.

Ages: 30 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with asthma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
A questionnaire for bronchial mucus hypersecretion | 1 year
  To design and validate a questionnaire to objectively assess the level of bronchial mucus hypersecretion

SECONDARY OUTCOMES:
Correlation of the results of the questionnaire with exacerbations | 1 year
  Perform a statistical analysis to determine the correlation of the results of the questionnaire with exacerbations
Correlation of the results of the questionnaire with FEV1 | 1 year
  Perform a statistical analysis to determine the correlation of the results of the questionnaire with FEV1
Correlation of the results of the questionnaire with ACT | 1 year
  Perform a statistical analysis to determine the correlation of the results of the questionnaire with FEV1

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Crespo-Lessmann, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau. Carrer Mas Casanovas 90., Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Fahy JV, Dickey BF. Airway mucus function and dysfunction. N Engl J Med. 2010 Dec 2;363(23):2233-47. doi: 10.1056/NEJMra0910061. No abstract available. PMID 21121836
- [Background] Rose MC, Voynow JA. Respiratory tract mucin genes and mucin glycoproteins in health and disease. Physiol Rev. 2006 Jan;86(1):245-78. doi: 10.1152/physrev.00010.2005. PMID 16371599
- [Background] Evans CM, Koo JS. Airway mucus: the good, the bad, the sticky. Pharmacol Ther. 2009 Mar;121(3):332-48. doi: 10.1016/j.pharmthera.2008.11.001. Epub 2008 Nov 18. PMID 19059283
- [Background] Walter MJ, Morton JD, Kajiwara N, Agapov E, Holtzman MJ. Viral induction of a chronic asthma phenotype and genetic segregation from the acute response. J Clin Invest. 2002 Jul;110(2):165-75. doi: 10.1172/JCI14345. PMID 12122108
- [Background] Lange P, Parner J, Vestbo J, Schnohr P, Jensen G. A 15-year follow-up study of ventilatory function in adults with asthma. N Engl J Med. 1998 Oct 22;339(17):1194-200. doi: 10.1056/NEJM199810223391703. PMID 9780339
- [Background] Aikawa T, Shimura S, Sasaki H, Ebina M, Takishima T. Marked goblet cell hyperplasia with mucus accumulation in the airways of patients who died of severe acute asthma attack. Chest. 1992 Apr;101(4):916-21. doi: 10.1378/chest.101.4.916. PMID 1555462
- [Background] Ordonez CL, Khashayar R, Wong HH, Ferrando R, Wu R, Hyde DM, Hotchkiss JA, Zhang Y, Novikov A, Dolganov G, Fahy JV. Mild and moderate asthma is associated with airway goblet cell hyperplasia and abnormalities in mucin gene expression. Am J Respir Crit Care Med. 2001 Feb;163(2):517-23. doi: 10.1164/ajrccm.163.2.2004039. PMID 11179133
- [Background] Martinez-Rivera C, Crespo A, Pinedo-Sierra C, Garcia-Rivero JL, Pallares-Sanmartin A, Marina-Malanda N, Pascual-Erquicia S, Padilla A, Mayoralas-Alises S, Plaza V, Lopez-Vina A, Picado C. Mucus hypersecretion in asthma is associated with rhinosinusitis, polyps and exacerbations. Respir Med. 2018 Feb;135:22-28. doi: 10.1016/j.rmed.2017.12.013. Epub 2018 Jan 3. PMID 29414449
- [Background] Carroll N, Elliot J, Morton A, James A. The structure of large and small airways in nonfatal and fatal asthma. Am Rev Respir Dis. 1993 Feb;147(2):405-10. doi: 10.1164/ajrccm/147.2.405. PMID 8430966
- [Background] Lopez-Vidriero MT, Reid L. Chemical markers of mucous and serum glycoproteins and their relation to viscosity in mucoid and purulent sputum from various hypersecretory diseases. Am Rev Respir Dis. 1978 Mar;117(3):465-77. doi: 10.1164/arrd.1978.117.3.465. PMID 629481
- [Background] Fleury Y, Dayem MA, Montagne JJ, Chaboisseau E, Le Caer JP, Nicolas P, Delfour A. Covalent structure, synthesis, and structure-function studies of mesentericin Y 105(37), a defensive peptide from gram-positive bacteria Leuconostoc mesenteroides. J Biol Chem. 1996 Jun 14;271(24):14421-9. doi: 10.1074/jbc.271.24.14421. PMID 8662868
- [Background] Crespo-Lessmann A, Plaza V; Consensus Group. Multidisciplinary consensus on sputum induction biosafety during the COVID-19 pandemic. Allergy. 2021 Aug;76(8):2407-2419. doi: 10.1111/all.14697. Epub 2021 Jan 19. PMID 33314245